CLINICAL TRIAL: NCT01569984
Title: An Open Label, Single-Centre, Phase II Study for Radiosensitization of AVASTIN® (Bevacizumab) With Stereotactic Body Radiotherapy (SBRT) for Colorectal Liver Metastasis (SBRT Avastin)
Brief Title: Radiosensitization of AVASTIN® (Bevacizumab) With Stereotactic Body Radiotherapy for Colorectal Liver Metastasis
Acronym: SBRT-Avastin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dr. Yoo-Joung Ko (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor-Investigator, Dr. Yoo-Joung Ko, Medical Oncoolgist, Sunnybrook Health Sciences Centre
Organization: Sunnybrook Health Sciences Centre (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OZM-032
Record Dates: First submitted 2012-03-30; First posted 2012-04-03 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-10

CONDITIONS: Colorectal Cancer.
Keywords: Colorectal
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Radiosurgery; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Avastin, SBRT (Experimental): 2 treatments of avastin followed by 6 treatments of SBRT every other day.
  Interventions: Radiation: Stereotactic body radiotherapy

INTERVENTIONS:
Radiation: Stereotactic body radiotherapy — Avastin 7.5 mg/kg IV x 2 doses 14 days apart
  Other Names: Bevacizumab

SUMMARY:
This is a single-centre, single-arm open-label proof-of-concept study to analyze the imaging (DCE-CT,CEUS and Quantitative US) effects of neoadjuvant bevacizumab and SBRT on colorectal metastases to the liver. Patients will receive 2 doses of bevacizumab 5mg/kg IV prior to SBRT. The second dose of bevacizumab will be given 2 weeks after the first dose of bevacizumab and within 48 hours of starting the first dose of SBRT. The SBRT prescription dose will be up to 60 Gy in 6 fractions, delivered on alternating weekdays for 2 weeks. Total SBRT dose will be determined by size of target lesion, liver sparing and organs-at-risk dose constraints. DCE-CT, CEUS and Quantitative US will be performed within 7 days prior to the first dose of bevacizumab, after the second dose of bevacizumab and within 7 days of completing SBRT.

DETAILED DESCRIPTION:
This is a single-centre, single-arm open-label proof-of-concept study to analyze the imaging (DCE-CT,CEUS and Quantitative US) effects of neoadjuvant bevacizumab and SBRT on colorectal metastases to the liver. Patients will receive 2 doses of bevacizumab 5mg/kg IV prior to SBRT. The second dose of bevacizumab will be given 2 weeks after the first dose of bevacizumab and within 48 hours of starting the first dose of SBRT. The SBRT prescription dose will be up to 60 Gy in 6 fractions, delivered on alternating weekdays for 2 weeks. Total SBRT dose will be determined by size of target lesion, liver sparing and organs-at-risk dose constraints. DCE-CT, CEUS and Quantitative US will be performed within 7 days prior to the first dose of bevacizumab, after the second dose of bevacizumab and within 7 days of completing SBRT.

ELIGIBILITY:
Inclusion Criteria:

1. Histological and/or cytological diagnosis of colorectal cancer with liver metastases confirmed on imaging scans
2. 1-3 liver metastatic lesions confirmed on imaging scans
3. Maximum size of target metastatic lesion is 6 cm or less
4. At least 700 cc of liver uninvolved by tumour
5. Previous liver resection, systemic therapy or local ablation therapy is allowed. Extrahepatic disease is allowed if maximum involved organs (including the liver) is 3 or less (i.e. oligometastases).
6. Child-Pugh's A liver function
7. Male or female: Age ≥ 18 years
8. Life expectancy > 3 months
9. ECOG PS < 2
10. Prior bevacizumab is permitted as long as last dose >28 days from registration
11. Laboratory Requirements - within 7 days prior to registration: Hematology

    * neutrophils ≥ 1.5 x 109/L
    * platelets ≥ 100 x 109/L
    * hemoglobin ≥ 90 g/L Biochemistry
    * bilirubin ≤ 1.5 x upper limit of normal
    * serum creatinine ≤ 1.5 x upper limit of normal
    * AST ≤ 3 x upper limit of normal (≤ 5 x if liver metastases present)
    * ALT ≤ 3 x upper limit of normal (≤ 5 x if liver metastases present)
    * INR ≤ 1.3 Urinalysis
    * Proteinuria ≤ grade 1 (by dipstick)
12. Patients are willing to provide informed consent.
13. Patients must be accessible for treatment and follow up. Patients registered on this trial must be treated and followed at the participating centre

Exclusion Criteria:

1. Major surgical procedure, open biopsy or significant traumatic injury within 28 days prior to registration (i.e. patients must have recovered to less than or equal to grade 1 from any major surgery), or anticipation of need for major surgical procedure during or within 7 weeks after chemo-radiotherapy.
2. Known to have clinical or radiological evidence of CNS metastases.
3. Patients with a past or current history (within last 2 years) of other malignancies, except for the indication under this study and curatively treated basal and squamous skin cancer or in-situ cancer of the cervix. Prior treatment of localized prostate cancer is permitted if treatment was greater than 5 years ago and the patient currently has no biochemical evidence of recurrence.
4. Active hepatitis (infectious or non-infectious)
5. Patients with known history or present encephalopathy
6. Gross clinically detectable ascites
7. Women of childbearing potential with a positive pregnancy test at baseline or lactating. Postmenopausal women must have been amenorrheic for at least 12 months to be considered of non childbearing potential. Females patients must not be pregnant or become pregnant during this study and for 6 months after the last dose of bevacizumab.
8. Sexually active males and females (of childbearing potential) unwilling to practice contraception during the study. Patients of childbearing potential must be willing to use a reliable method of birth control. i.e.:double barrier method, oral contraceptive, implant, dermal contraception, long-term injectable contraceptive, intrauterine device or tubal ligation during the study.
9. Prior radiotherapy to the right upper quadrant of the liver
10. Known hypersensitivity reaction to bevacizumab
11. Known hypersensitivity to Chinese hamster ovary cell products or other recombinant human or humanised antibodies
12. Uncontrolled hypertension, defined as SBP > 150/100 on more than one occasion that does not respond to therapy with antihypertensive agents or being treated with more than 2 anti-hypertensive medications.
13. Any other serious intercurrent illness such as cardiovascular disease, HIV or any neurological disease.
14. Patients taking other approved or investigational drug/anticancer treatment (other than ongoing androgen ablation and oral prednisone which are permitted) during the study period, including chemotherapy, biological response modifiers, immunotherapy, surgery or radiotherapy.
15. Patients concurrently participating in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2012-03; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Tumor perfusion | day 24
  Tumor perfusion as measured by DCE-CT

SECONDARY OUTCOMES:
Blood flow | Day 24
  Contrast Enhanced Ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Yoo-Joung Ko, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada